CLINICAL TRIAL: NCT06900140
Title: Adjunctive Methylene BLUe in Septic SHock: a Pilot Randomized Controlled Trial
Brief Title: Adjunctive Methylene Blue in Septic Shock
Acronym: BLUSH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Shannon M. Fernando (Other)
Responsible Party: Sponsor-Investigator, Dr. Shannon M. Fernando, Principal Investigator, Lakeridge Health
Organization: Lakeridge Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHICU123
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Septic Shock
Keywords: Septic shock; Methylene blue
MeSH Terms: conditions — Shock, Septic | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene Blue (Experimental): Methylene Blue infusion: 0.5 mg/kg/hr for 6 hours daily (up to 3 days total).
  Interventions: Drug: Methylene Blue
- Usual Care (Active Comparator): Usual guideline-directed care for adult septic shock.
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Methylene Blue — Continuous methylene blue infusion at a fixed dose of 0.50 mg/kg/hour (diluted in 500 mL of dextrose 5% in water) over 6 hours once daily, for a total of up to 3 doses.
  Arms: Methylene Blue
Other: Usual Care — Usual guideline-directed care for adult septic shock.
  Arms: Usual Care

SUMMARY:
Adjunctive Methylene BLUe in Septic SHock (BLUSH) is a single centre concealed-allocation parallel-group open-label randomized controlled pilot trial to ascertain the feasibility of a trial evaluating the efficacy and safety of adjunctive methylene blue infusion compared to usual care on outcomes of adult patients admitted to the intensive care unit with septic shock.

DETAILED DESCRIPTION:
BACKGROUND: Septic shock remains an important cause of morbidity and mortality worldwide, and disproportionately affects low- and middle-income countries. The current standard of care in the treatment of septic shock is limited to antimicrobials and supportive care such as intravenous fluids, vasopressors, mechanical ventilation, and renal replacement therapy. Existing data from small randomized controlled trials suggests that methylene blue may be efficacious in reducing vasopressor exposure and mortality in patients with septic shock. Methylene blue is an inexpensive and readily available therapy which, if proven effective, could be used worldwide and drastically change outcomes in high- and low-income settings alike.

OBJECTIVES: Pilot trial to determine the feasibility of a large, open-label, multicentre randomized trial evaluating the efficacy and safety of intravenous methylene blue infusion, as compared to usual care, in adult patients with septic shock in the intensive care unit (ICU).

METHODS: Patients will be randomly assigned to methylene blue infusion (intravenous, dissolved in dextrose 5% in water, run at 0.5 mg/kg/hr over 6 hours daily) up to 3 days total, or usual care for septic shock. Study personnel at the clinical sites will document the composite of death or persistent organ dysfunction at day 28. Daily assessments will occur for organ function and vasopressor exposure. The trial will be conducted in two adult intensive care units at Lakeridge Health.

RELEVANCE: The BLUSH trial will test the feasibility of conducting a large randomized trial to evaluate the efficacy and safety of methylene blue in adult patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years of age) admitted to the ICU
2. Diagnosed with septic shock (as per the Sepsis-3 Criteria): Suspected infection (i.e. initiation of antimicrobial therapy), coupled with initiation of vasopressor therapy to target a mean arterial pressure (MAP) > 65 mmHg (or as prescribed by the treating clinician), after adequate fluid resuscitation (as per treating clinician).
3. Minimal norepinephrine dose of 0.1 mcg/kg/min for a minimum of 2 hours at the time of enrollment (i.e., the time of randomization).

Exclusion Criteria:

1. > 48 hours since initiation of norepinephrine
2. > 48 hours since admission to ICU
3. Anticipation of discontinuation of vasopressors in < 24 hours
4. Pregnancy **Women of childbearing age (<50 years) should have a urine or beta hCG performed prior to enrolment
5. Plan for withdrawal of life support
6. Concurrent hemorrhagic, obstructive, or hypovolemic shock
7. Major burn injury (>10% total body surface area)
8. Known Personal or familial history of glucose-6-phophate dehydrogenase deficiency
9. Known Allergy to methylene blue, phenothiazines, or food dyes
10. Known recent intake of selective serotonin re-uptake inhibitors (21 days for norfluoxetine, and 14 days for any other SSRI).
11. Currently receiving linezolid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Enrolment/Recruitment Rate | Enrolment
  The investigators define a successful recruitment rate of 1 patient per centre per month over the duration of the trial. The recruitment will be reviewed weekly and the screening logs will be reviewed monthly. This will be done to ensure that enrolment is being maximized and that any barriers are being addressed. A recruitment metric will be measured and interpreted at the end of the trial. Excluded patients and eligible non-randomized patients will be reviewed to determine whether any modifications to the protocol may be warranted, or to address implementation challenges. Barriers to enrolment will be discussed and strategies to improve enrolment will be operationalized, if needed.
Consent Rate | Enrolment
  The investigators will define >50% consent rate as successful. This will be calculated as the overall proportion of patients/substitute decisions makers (SDMs) who consented to the trial out of everyone who was approached. If a patient or SDM chooses to withdraw from the study but allows for the data that had been collected up until that point to be used for analysis, they will still be counted as providing consent. Reasons for withdrawal will be recorded. The consent rate will be reviewed weekly and any barriers to consent that are identified will be addressed to improve the consent process.
Protocol Adherence | Enrolment
  The investigators will define ≥80% protocol adherence as successful. The adherence will be calculated as the number of patients who received allocated therapy per eligible study day over all the eligible study intervention days across enrolled patients. Each enrolled patient will contribute 3 eligible study intervention days unless they meet discontinuation criteria (e.g., stopped vasopressors). The research coordinator will review the chart to determine the actual compliance, and document all the reasons for non-compliance of both the control and experimental arms of the study. Furthermore, the study drug being discontinued and then re-started in a study patient would also not be deemed a protocol violation. Adherence will also be reviewed monthly and the reasons for compliance failure will be investigated and recorded as a protocol violation. Further behavioural strategies will be employed to improve adherence, if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Fernando, MD, Principal Investigator — Lakeridge Health
Locations (1):
- Lakeridge Health, Oshawa, Ontario, Canada